CLINICAL TRIAL: NCT02316249
Title: Vaginal Creams for Reduction of Vaginal Discharge and Erosion in Patients Using Ring With Support or Gellhorn Pessaries to Reduce Pelvic Organ Prolapse
Brief Title: Vaginal Creams to Reduce Vaginal Erosion in Pessary Users
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: the study was not feasible
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Lawrence Lind, Principal Investigator, Northwell Health
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: NSHS-P001
Record Dates: First submitted 2014-12-10; First posted 2014-12-12 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Atrophy of Vagina; Vaginal Ulceration; Vaginitis
Keywords: pelvic organ prolapse; Atrophy of Vagina; Gellhorn pessary; Ring with support pessary; Estrace cream; vaginitis with pessary; vaginal ulceration with pessary; vaginal erosion with pessary; pessary complications; vaginal bleeding with pessary
MeSH Terms: conditions — Vaginitis; Pelvic Organ Prolapse | interventions — Estradiol; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gellhorn Pessary (Active Comparator): Patients who are fitted with a Gellhorn pessary for reduction of pelvic organ prolapse. Patients will then be randomized based on pessary to either Estradiol vaginal cream or Placebo vaginal cream. Patients will be instructed to digitally apply 0.5mg of cream inside vagina every night for 2 weeks. After 2 weeks they will switch to 2 nights weekly.
  Interventions: Drug: Estradiol; Other: placebo
- Ring with Support Pessary (Active Comparator): Patients who are fitted with a Ring with Support Pessary for reduction of pelvic organ prolapse. Patients will then be randomized based on pessary to either Estradiol vaginal cream or Placebo vaginal cream. Patients will be instructed to digitally apply 0.5mg of cream inside vagina every night for 2 weeks. After 2 weeks they will switch to 2 nights weekly.
  Interventions: Drug: Estradiol; Other: placebo

INTERVENTIONS:
Drug: Estradiol — Patients will be instructed to digitally apply 0.5mg of cream inside vagina every night for 2 weeks. After 2 weeks they will switch to 2 nights weekly.
  Other Names: Estrace
Other: placebo — Patients will be instructed to digitally apply 0.5mg of cream inside vagina every night for 2 weeks. After 2 weeks they will switch to 2 nights weekly.
  Other Names: A hormone free base for vaginal creams

SUMMARY:
To compare the use of Estrace ® vaginal cream against a placebo vaginal cream in reducing symptomatic vaginal discharge and vaginal erosion in patients who are using the Gellhorn or Ring with support pessaries.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is a health concern for millions of women worldwide. Patients have a variety of symptoms from POP including: vaginal bulging, vaginal pressure, constipation and urinary incontinence (1). It is estimated that the lifetime risk of undergoing surgery for prolapse or incontinence is 11%. The lifetime risk for recurrence of POP after surgery is 10-20% (2). Treatment options for POP include kegel exercises, pessaries or surgical management. Due to lifestyle, timing or inability to undergo surgery secondary to medical comorbidities the pessary can be a very reasonable alternative to surgical management of POP.

There are two categories of pessaries: support and space occupying. Support pessaries are usually recommended for early stage of prolapse with adequate perineal support and include the ring pessary, Gehrung, Hodge and Shaatz. While space-occupying pessaries such as the Donut, Gellhorn, Cube and Inflataball are used for advanced stage prolapse with less perineal support and a wide genital hiatus (3). As the ring and the Gellhorn pessary are the most commonly used pessaries and can be inserted for all stages of prolapse, our study will focus on the use of the ring with support and the Gellhorn for treatment of POP (4).

After menopause, estrogen levels decline. This may allow postmenopausal vaginal pH to increase to the range of 5.0-7.5. At these higher pH levels, lactobacillus survival is hindered, and vaginal colonization by other bacterial species predisposes women to symptomatic vaginitis (5). Discontinuation of pessary use is often due to discomfort, expulsion, urinary retention bothersome vaginal discharge and vaginal erosion (6). Common complications with pessary use are erosions (8.9%), or vaginal infections (2.5%) (7). Some studies have shown an erosion rate as high as 21% (6). Patients often complain of vaginal discharge with pessary use that is malodorous and bothersome. Local estrogen can help to restore the vaginal pH and help reduce vaginal discharge. The moisturizing properties of vaginal lubricants and creams may help reduce vaginal erosion in pessary users. We would like to compare Estrace ® to a placebo. The placebo will be the hormone replacement therapy (HRT) base cream in Estrace ® without the estradiol.

No randomized control trials (RCT) have been performed showing if application of local hormone (Estrace) is superior to application of local nonhormonal vaginal cream for reduction of the bothersome symptom of vaginal discharge and subsequently erosion. We would like to compare vaginal estrogen against placebo as a mechanism to prevent bothersome discharge and prevention of vaginal erosion in women fitted with pessaries for pelvic organ prolapse.

Study Population In general, the study population will be patients of the Urogynecology practice of North Shore-Long Island Jewish Health System who present to the clinic for their initial pessary fitting. Patients will be fitted with either a ring with support or Gellhorn pessary and will return at intervals of 2, 6 and 12 weeks for follow up.

All subjects over 18 yrs of age will be screened for eligibility relative to the patient inclusion and exclusion criteria. If a patient is eligible to enroll in the study, the nature and purpose of the study will be explained to the subject with a witness present. The subject will review and sign the written Informed Consent Form indicating informed and voluntary participation in the study. A copy of the consent form including all risks and benefits to the research subjects is attached as a separate document.

Recruitment for the study will be done via direct contact from our patient population. If a subject is found to be eligible to participate, an approved study investigator will approach her during her scheduled initial pessary visit. No form of advertisement will be used. The recruitment methods used will provide equitable selection of subjects.

After determination of eligibility based on inclusion/exclusion criteria the patient will be consented for the study related procedures. The subject must consent to participate and sign the specific Institutional Review Board approved Informed Consent Form prior to the conduct of the study specific procedure. Patient may be consented in the clinic for the department of urogynecology.

New patients who present for their initial pessary fitting will have the appropriate sized ring with support or Gellhorn pessary placed as per standard of care. The patient will return for her 2 week follow up visit as per standard of care.

If no change in pessary is indicated the patient will be approached for participation in the study. If she agrees to participate, she will be randomized to use estrogen cream (Estrace) or placebo stratified on type of pessary.

Estrace contains 0.1 mg estradiol per gram of cream. The recommended dosing is 2-4 grams daily for 1-2 weeks with a gradual reduction to half the initial dose over 1-2 weeks, and then 1 gram 1-3 times weekly for maintenance.

Participants will be provided with the medication in prepackaged 0.5cc syringe. Either digitally or by using the syringe, she will then place 1cm distal to the introitus. This technique will be reviewed with the participant and she will also have to demonstrate correct application. She will use the cream nightly for 1 week then reduce the dose to 2 times weekly for maintenance. Participants will use the cream nightly for 1 week then twice weekly at night.

The patient will be given a 3 month supply of the vaginal cream that she is randomized to. We will preload syringes with 0.5cc of either estrace or placebo cream. These will be randomized by a non-blinded study personnel.

Study participants will return for follow-up appointments at 2 weeks, 6 weeks, 12 weeks and 6 months. Participants will also be expected to return all syringes that she has used prior to the scheduled visit. This will aid in our assessment of patient compliance with suggested use of medication and also ensure that correct disposal of the vaginal cream.

As per standard of care, a vaginal culture will be obtained at any visit if the patient complains of a bothersome, malodorous discharge. In addition to the vaginal culture, patients who report a malodorous discharge will undergo saline irrigation at time of visit and examination of vaginal tissue for erosion. If no vaginal erosion present the pessary will be replaced and the patient will be instructed to continue the previously prescribed regimen of 3 times weekly application of vaginal cream. If vaginal erosion is noted, the pessary will be left out for 3 weeks and the patient will be instructed to use the vaginal cream daily for 3 weeks. The patient will then return to the office after 3 weeks for a vaginal exam and replacement of pessary upon resolution of vaginal erosion.

We will assess for atrophy, erosion, vaginal discharge and obtain a vaginal culture if clinically applicable. Questionnaires will be completed at baseline, 12 week and 6 month follow-up visits and include: Pelvic Floor Distress Inventory (PFDI), Pelvic Floor Impact Questionnaire (PFIQ). We will assess patient satisfaction for use of pessary at each follow-up using a Liekhart scale. Patients with bothersome vaginal discharge will use a VAS scale with a rating of with a 10cm linear continuum in which 0 represents very bothersome and 10 represents not at all bothersome. Vaginal erosion will be clinically described as minimal, moderate or severe.

This research may not benefit study participants directly. However, knowledge gained from this study may help physicians and patients in the future with regard to the best treatment to reduce vaginal discharge and vaginal erosion in pessary users.

Potential risks for this study outside of the risks associated with pessary use are minimal. Complications with pessary use include: vaginal erosion, urinary retention, urinary incontinence and discomfort. These complications will be reviewed with the patient prior to insertion of pessary. Potential risks encountered when using vaginal estrogen are low. Estrace contains 0.1 mg estradiol per gram of cream. The recommended dosing is 2-4 g daily for 1-2 weeks, a gradual reduction to half the initial dose over 1-2 weeks, and then 1 g 1-3 times weekly for maintenance. Our patients will be using half the recommended daily dose for maintenance and at the most, 1/4th the recommended dose for priming the atrophic tissue.

We are also reducing an additional minimal risk associated with local vaginal estrogen in our exclusion criteria.

If a participant reports that she has not used the cream or has returned the syringes unused, she will be removed from the study for lack of compliance. Study participants will also be removed from the study if they develop or have a new diagnosis of any conditions that are listed in the exclusion criteria. Finally, they will be removed if any allergic reactions/adverse events occur from the use of Estrace or placebo. There will be no replacement procedure for study participants if they are withdrawn. No actions will follow or are warranted after study participant removal.

This is a double-blinded randomized control trial of subjects with pelvic organ prolapse who, after counseling at their initial visit, opt for treatment with a vaginal pessary. Patients who have a Gellhorn or Ring with support pessary placed with then be randomized to one of two arms for application of a local vaginal cream: estrogen or placebo. The object of the study is to compare the incidence of vaginal discharge and vaginal erosion in each study arm. We will also compare subjective measures including quality of life and satisfaction with their treatment plan.

Our Primary Objective is to compare the use of Estrace® or placebo in reducing symptomatic vaginal discharge and vaginal erosion in patients using Gellhorn or Ring pessaries.

Prior to randomization subjects will be stratified according to type of pessary (Gellhorn or Ring). Within a stratum, subjects will be randomly assigned in a 1:1 ratio to Estrace® or placebo.

The Biostatistics Unit will develop a computer-generated randomization list that utilizes a permuted block design, and will develop and implement a well documented double-blind randomization procedure.

Intention-to-treat (ITT):

Data collected will be analyzed according to the ITT principle. The ITT population will be all patients randomized, regardless of whether or not the study cream was applied. All patients will be analyzed in the group to which they were randomized (even if they are switched over to another cream.)

Patients will be assessed for study data at baseline (once the pessary is placed successfully, week 0), 6, 12, and 24 weeks.

Descriptive statistics (means ± standard deviations or medians and interquartile range [25th percentile, 75th percentile] for continuous data; frequencies and percentages for categorical data) will be calculated for subjects on demographic and clinical characteristics as well as outcomes observed at the end of the trial.

The two groups will be compared for categorical variables using the chi-square test or Fisher's exact test, as deemed appropriate. The two-sample t-test or Mann-Whitney test will be used to compare the two groups for continuous data.

Separate repeated measures analysis of variance (RMANOVA) models using a mixed models approach will be used to compare the two treatment arms with respect to their vaginal discharge, POP-Q staging , PFDI, and PFIQ trajectories from baseline to 24 weeks. Each model will include the main effects of treatment arm (Estrace® or placebo) and time (0, 12, and 24 weeks), as well as the treatment x time interaction. If an interaction between group and time is not found to be statistically significant, only the main effects of treatment group and time will be analyzed. For all analyses, the standard assumptions of Gaussian residuals and quality of variance will be tested. If the standard assumptions are not met, a transformation will be performed.

A result will be considered statistically significant at the p<0.05 level of significance. All analyses will be performed using SAS version 9.3 (SAS Institute, Cary, NC).

The proposed sample size for this double-blind randomized control trial is n=246 subjects (n=123 per arm).

Based on data published by Manchana , 21% of symptomatic pelvic organ prolapse patients fitted successfully with a pessary had vaginal erosion. Let us assume a 60% reduction from this estimate (21% to 8.4%) after using Estrace®. A two group χ2 test with a 0.05 two-sided significance level will have 80% power to detect the difference between a vaginal erosion rate for the placebo group = 0.21 and a vaginal erosion rate of the Estrace® group = 0.084 when the sample size in each group is 123.

Our study limitations are that our primary outcome is a subjective assessment of vaginal discharge and vaginal erosion. Our population is an older, postmenopausal population and therefore may be more susceptible to vaginal erosion. Patient compliance to use of the vaginal cream 2 times weekly is also another limitation as this is a patient directed cannot be controlled, however we will try to reduce this limitation by requiring that patients bring their used syringes back to the office.

The PI will monitor data, with emphasis on data integrity and patient welfare concerns including: recommendations concerning continuation or conclusion of the study, protection of the confidentiality of the trial data and the results of monitoring, review of data and study quality.

Any adverse events, unanticipated problems, and protocol deviations will be reported to the Institutional Review Board as per North Shore-Long Island Jewish Health System policy.

Confidentiality will be maintained by using patient identification numbers instead of names. Original documents including consent forms that contain subjects' PHI, as well as questionnaires, will be stored in a locked cabinet within the office of Urogynecology, 865 Northern Blvd., Suite 202, Great Neck, New York 11021. These documents will be kept separately from any de-identified research data that will be stored electronically as mentioned below. Institutional Review Board approved investigators will be the only individuals with access to research data that contains PHI. Any documents that contain subjects' PHI will be accessible on the North Shore-Long Island Jewish Health System network server through a password protected computer document/database. These documents are separated from any de-identified research data files. Institutional Review Board approved investigators will be the only individuals with access to research data that contains PHI. De-identified data research files will be stored on the network server.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Female gender
* >/= Stage II pelvic organ prolapse
* Clinical diagnosis of pelvic organ prolapse and desiring non-surgical management with pessary
* Ability to provide informed consent and complete all study requirements

Exclusion Criteria:

* Life expectancy < 12 months
* Current pregnancy
* Patients will undergo a urine pregnancy test
* Already using vaginal estrogen
* Limited manual dexterity
* History of vaginal erosion with prior pessary use
* All patients with a past or present diagnosis of Breast cancer
* Patients with any pathology of the female reproductive organs
* Patients with undiagnosed abnormal genital bleeding
* Patients with known or suspected estrogen-dependent neoplasia
* Active deep vein thrombosis, pulmonary embolism or history of these conditions
* Active or recent (within last year) arterial thromboembolic disease
* Patients with liver dysfunction or disease
* Patients with known hypersensitivity to Estrace's ingredients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Vaginal erosion | 6 months
  To assess erosion/ulceration of vaginal tissue in patients using a Ring with support or Gellhorn Pessary for treatment of >/= Stage II Pelvic Organ Prolapse

SECONDARY OUTCOMES:
Reason for Discontinuation of pessary based on style of pessary | 6 months
  We will record patient& reason for discontinuation of pessary. A common reason for discontinuation is vaginal discharge.
Patient satisfaction with Pessary (Pelvic Floor Distress Inventory (PFDI) | 6 months
  Using the Pelvic Floor Distress Inventory (PFDI) Questionnaire and the Pelvic Floor Impact Questionnaire. We will assess patient satisfaction with reduction of prolapse via pessary and symptomatic improvement
vaginal discharge/vaginitis | 6 months
  To document whether the patient has a bothersome vaginal discharge. If so, we will perform a wet mount and/or vaginal culture for assessment and treatment of vaginitis.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lind, MD, Principal Investigator — Hofstra North Shore
Locations (1):
- Division of Urogynecology North Shore-LIJ School of Medicine, Great Neck, New York, United States